CLINICAL TRIAL: NCT00544882
Title: A Prospective, Multicenter, Randomized, Double-Blind Study to Evaluate Hormone Patterns and Ovarian Follicular Activity With the Oral Contraceptive Regimen DR-1021
Brief Title: A Study to Evaluate Hormone Patterns and Ovarian Follicular Activity With DR-1021
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-DSG-302
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Desogestrel; Oviol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DR-1021 (Experimental): After randomization, participants received DR-1021 consisting of 150 μg desogestrel (DSG)/20 μg ethinyl estradiol (EE) administered orally as a combination tablet once daily for 21 days followed by EE 10 μg tablet once daily for 7 days (Cycle 2). Participants who completed Cycle 2 then received Kariva, consisting of 150 μg DSG/20 μg EE administered orally as a combination tablet taken once daily for 21 days followed by placebo tablet once daily for 2 days followed by 10 μg EE taken once daily for 5 days (Cycle 3).
  Interventions: Drug: DR-1021; Drug: Kariva®
- Mircette (Active Comparator): After randomization, participants received Mircette consisting of 150 μg desogestrel (DSG)/20 μg ethinyl estradiol (EE) administered orally as a combination tablet once daily for 21 days followed by placebo tablet once daily for 2 days followed by 10 μg EE tablet once daily for 5 days (Cycle 2). Participants who completed Cycle 2 then received Kariva, consisting of 150 μg DSG/20 μg EE administered orally as a combination tablet taken once daily for 21 days followed by placebo tablet once daily for 2 days followed by 10 μg EE taken once daily for 5 days (Cycle 3).
  Interventions: Drug: Mircette®; Drug: Kariva®

INTERVENTIONS:
Drug: DR-1021 — Twenty-one 150 μg desogestrel/20 μg ethinyl estradiol (EE) combination tablets plus seven 10 μg EE tablets.
  Other Names: desogestrel/ethinyl estradiol
  Arms: DR-1021
Drug: Mircette® — Twenty-one 150 μg desogestrel/20 μg ethinyl estradiol (EE) combination tablets plus two placebo tablets plus five 10 μg EE tablets.
  Other Names: desogestrel/ethinyl estradiol
  Arms: Mircette
Drug: Kariva® — Twenty-one 150 μg desogestrel/20 μg ethinyl estradiol (EE) combination tablets plus two placebo tablets plus five 10 μg EE tablets.
  Other Names: desogestrel/ethinyl estradiol

SUMMARY:
This is a multi-center study to evaluate hormone levels with the oral contraceptive regimen DR-1021.

DETAILED DESCRIPTION:
Female volunteers, aged 18-35 years old who met all Inclusion and no Exclusion Criteria, were enrolled in this study. All participants were current users of a standard 21/7 oral contraceptive regimen (21 days of combination progestin/estrogen followed by 7 days placebo) and had completed at least one 28-day cycle prior to beginning the Cycle 1 baseline cycle. After completing screening, all enrolled participants continued to receive the same regimen of 150 μg DSG /20 μg EE combination pills once daily for 21 days followed by placebo once daily for 7 days during Cycle 1 (the Run-In phase). Following completion of Cycle 1, participants were randomly assigned to receive either DR-1021 or Mircette during Cycle 2. All participants who completed Cycle 2 were to receive Kariva during Cycle 3; however, participants were only followed for the first 21 days of this 28-day regimen, after which they were considered study completers.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Weight <200 lbs
* Currently taking or willing to be treated with an oral contraceptive with a standard 21/7 regimen for one cycle prior to starting Study Cycle 1
* Others as dictated by protocol

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Breast feeding
* Smoking > 10 cigarettes per day
* Use of drugs that require simultaneous use of contraceptives (e.g., isotretinoin [Accutane])
* Others as dictated by protocol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2007-10-31 (Actual); Primary Completion 2008-03-31 (Actual); Study Completion 2008-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (4):
- United States (4):
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female volunteers, aged 18-35 years old who were current users of a standard 21/7 oral contraceptive regimen (21 days of combination progestin/estrogen followed by 7 days placebo) were enrolled at 4 investigative sites in the United States.
Pre-assignment Details: 67 women were screened for participation in this study; 61 were enrolled and took at least 1 dose of their current regimen of oral contraceptive in Cycle 1 (the Run-in Cycle). Of the 61 enrolled, 3 participants discontinued the study prior to completing the Run-in Cycle and were therefore not randomly assigned to study drug in Cycle 2.
Groups:
- Run-In Cycle - All Enrolled: After completing screening, all enrolled participants received the same regimen of 150 μg Desogestrel (DSG) /20 μg Ethinyl Estradiol (EE) combination pills once daily for 21 days followed by placebo once daily for 7 days during Cycle 1.
Period: Cycle 1: Run-in Cycle
Arm/Group | Run-In Cycle - All Enrolled | DR-1021 | Mircette
Started | 61 | 0 | 0
Completed | 58 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Cycle 2: Randomized Treatment Cycle
Arm/Group | Run-In Cycle - All Enrolled | DR-1021 | Mircette
Started | 0 | 29 | 29
Treated | 0 | 28 (One participant withdrew prior to treatment) | 28 (One participant was dropped from the study due to noncompliance prior to treatment.)
Completed | 0 | 28 | 28
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Noncompliance | 0 | 0 | 1
Period: Cycle 3: Follow-up
Arm/Group | Run-In Cycle - All Enrolled | DR-1021 | Mircette
Started | 0 | 28 | 28
Completed | 0 | 26 (Completed 21 days of Cycle 3) | 28 (Completed 21 days of Cycle 3)
Not Completed | 0 | 2 | 0
Not completed — Noncompliance | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) cohort consisted of all randomized participants who took at least one dose of randomized study medication and had at least one post-baseline efficacy measurement for at least one of the primary efficacy endpoints (FSH, inhibin-B, or estradiol).
Groups:
- Total: Total of all reporting groups
Arm/Group | DR-1021 | Mircette | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (4.68) | 28.0 (4.38) | 27.7 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 4 | 6 | 10
  Asian | 2 | 0 | 2
  Caucasian | 20 | 20 | 40
  Hispanic | 1 | 1 | 2
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Serum Estradiol Levels by Cycle Day
Description: Levels of estradiol were measured throughout the study from blood samples.
Time Frame: Cycle 2, Day 2 (Baseline), and Days 4, 6, 19-20, 23, 24, 25, 27, 28, Cycle 3, Days 2, 4 and 6.
Population: Intent-to-treat population with available data at each time point (as indicated by n).
Measure: Median (Full Range); unit: pg/mL
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
pg/mL
  Cycle 2 - Day 2 (n=28, 28) | 47.00 [15.0 to 361.0] | 51.50 [6.0 to 322.0]
  Cycle 2 - Day 4 (n=28, 28) | 62.50 [1.0 to 613.0] | 34.50 [1.0 to 423.0]
  Cycle 2 - Day 6 (n=27, 27) | 43.00 [1.0 to 579.0] | 29.00 [1.0 to 274.0]
  Cycle 2 - Days 19-20 (n=26, 28) | 19.00 [1.0 to 152.0] | 20.50 [1.0 to 327.0]
  Cycle 2 - Day 23 (n=27, 28) | 24.00 [1.0 to 204.0] | 19.00 [1.0 to 159.0]
  Cycle 2 - Day 24 (n=25, 28) | 25.00 [1.0 to 289.0] | 26.50 [1.0 to 169.0]
  Cycle 2 - Day 25 (n=27, 28) | 24.00 [1.0 to 169.0] | 26.00 [1.0 to 225.0]
  Cycle 2 - Day 27 (n=25, 28) | 30.00 [1.0 to 233.0] | 20.00 [1.0 to 213.0]
  Cycle 2 - Day 28 (n=26, 28) | 36.00 [1.0 to 284.0] | 27.50 [1.0 to 332.0]
  Cycle 3 - Day 2 (n=27, 28) | 34.00 [1.0 to 425.0] | 43.00 [3.0 to 217.0]
  Cycle 3 - Day 4 (n=27, 27) | 66.00 [1.0 to 440.0] | 27.00 [1.0 to 295.0]
  Cycle 3 - Day 6 (n=24, 26) | 28.50 [1.0 to 277.0] | 32.00 [3.0 to 197.0]
Statistical Analysis 1: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 2 time point. p-values < 0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.6346, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 4 time point; Test type: Superiority or Other; p = 0.2757, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 6 time point; Test type: Superiority or Other; p = 0.1321, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Days 19-20 time point; Test type: Superiority or Other; p = 0.5543, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 23 time point; Test type: Superiority or Other; p = 0.3940, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 24 time point; Test type: Superiority or Other; p = 0.7891, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 25 time point; Test type: Superiority or Other; p = 0.4829, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 27 time point; Test type: Superiority or Other; p = 0.4526, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 28 time point; Test type: Superiority or Other; p = 0.2485, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 2 time point; Test type: Superiority or Other; p = 0.6252, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 4 time point; Test type: Superiority or Other; p = 0.4003, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 6 time point; Test type: Superiority or Other; p = 0.8841, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage of Follicles Greater Than 5 mm in Diameter
Description: Ovarian follicles were measured by trans-vaginal ultrasound. The size of the 3 largest follicles was documented for each participant, and the percentage of follicles greater than 5 mm in diameter was calculated based on the total number follicles present (indicated by n for each time point).
Time Frame: Cycle 1, Days 11, 19-20, 23, 25, 27, Cycle 2, Days 4, 11, 19-20, 23, 25, 27, Cycle 3, Day 4.
Population: Intent-to-treat
Measure: Number; unit: percentage of follicles
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
percentage of follicles
  Cycle 1 - Day 11 (n=63, 48) | 30.2 | 29.2
  Cycle 1 - Day 19-20 (n= 47, 94) | 29.8 | 27.7
  Cycle 1 - Day 23 (n= 30, 76) | 50.0 | 26.3
  Cycle 1 - Day 25 (n= 85, 106) | 32.9 | 31.1
  Cycle 1 - Day 27 (n=135, 145) | 29.6 | 35.2
  Cycle 2 - Day 4 (n=154, 156) | 35.1 | 31.4
  Cycle 2 - Day 11 (n=76, 54) | 27.6 | 31.5
  Cycle 2 - Days 19-20 (n=143, 148) | 17.5 | 18.9
  Cycle 2 - Day 23 (n=91, 62) | 24.2 | 24.2
  Cycle 2 - Day 25 (n=69, 80) | 30.4 | 18.8
  Cycle 2 - Day 27 (n=94, 132) | 23.4 | 20.5
  Cycle 3 - Day 4 (n=138, 117) | 25.4 | 27.4

3. Primary Outcome: Serum Follicle Stimulating Hormone (FSH) Levels by Cycle Day
Description: Levels of follicle stimulating hormone were measured throughout the study from blood samples.
Time Frame: Cycle 2, Day 2 (Baseline), and Days 4, 6, 19-20, 23, 24, 25, 27, 28, Cycle 3, Days 2, 4 and 6.
Population: Intent-to-treat population with available data at each time point (as indicated by n).
Measure: Median (Full Range); unit: mIU/mL
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
mIU/mL
  Cycle 2 - Day 2 (n=28, 28) | 4.00 [2.3 to 9.7] | 4.00 [1.2 to 7.1]
  Cycle 2 - Day 4 (n=28, 28) | 3.55 [1.2 to 9.5] | 3.70 [0.9 to 28.8]
  Cycle 2 - Day 6 (n=28, 27) | 3.70 [0.4 to 8.5] | 3.50 [0.2 to 14.9]
  Cycle 2 - Days 19-20 (n=26, 28) | 1.45 [0.2 to 5.7] | 1.55 [0.2 to 8.1]
  Cycle 2 - Day 23 (n=27, 28) | 2.70 [0.2 to 6.3] | 2.35 [0.2 to 6.3]
  Cycle 2 - Day 24 (n=25, 28) | 2.80 [0.2 to 8.0] | 3.70 [0.2 to 8.4]
  Cycle 2 - Day 25 (n=27, 28) | 2.90 [0.2 to 8.0] | 3.90 [0.2 to 11.3]
  Cycle 2 - Day 27 (n=25, 28) | 3.70 [0.2 to 9.6] | 3.90 [0.3 to 8.3]
  Cycle 2 - Day 28 (n=26, 28) | 5.05 [0.2 to 11.0] | 4.70 [0.4 to 25.8]
  Cycle 3 - Day 2 (n=27, 28) | 4.90 [0.2 to 9.8] | 4.05 [0.2 to 10.2]
  Cycle 3 - Day 4 (n=27, 28) | 3.70 [0.2 to 8.0] | 3.60 [0.2 to 8.1]
  Cycle 3 - Day 6 (n=24, 26) | 2.50 [0.6 to 7.1] | 2.50 [0.2 to 8.8]
Statistical Analysis 1: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 2 time point. p-values < 0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.8892, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 4 time point; Test type: Superiority or Other; p = 0.7678, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 6 time point; Test type: Superiority or Other; p = 0.5782, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Days 19-20 time point; Test type: Superiority or Other; p = 0.8083, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 23 time point; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 24 time point; Test type: Superiority or Other; p = 0.4122, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 25 time point; Test type: Superiority or Other; p = 0.6675, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 27 time point; Test type: Superiority or Other; p = 0.8445, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 28 time point; Test type: Superiority or Other; p = 0.3772, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 2 time point; Test type: Superiority or Other; p = 0.1918, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 4 time point; Test type: Superiority or Other; p = 0.6675, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 6 time point; Test type: Superiority or Other; p = 0.9226, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Serum Inhibin-B Levels by Cycle Day
Description: Levels of inhibin-B were measured throughout the study from blood samples.
Time Frame: Cycle 2, Day 2 (Baseline), and Days 4, 6, 19-20, 23, 24, 25, 27, 28, Cycle 3, Days 2, 4 and 6.
Population: Intent-to-treat population with available data at each time point (as indicated by n).
Measure: Median (Full Range); unit: pg/mL
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
pg/mL
  Cycle 2 - Day 2 (n=28, 28) | 92.30 [3.5 to 157.9] | 99.00 [37.0 to 460.7]
  Cycle 2 - Day 4 (n=28, 28) | 42.80 [13.3 to 128.9] | 64.45 [15.9 to 197.0]
  Cycle 2 - Day 6 (n=28, 27) | 46.35 [3.5 to 186.9] | 41.20 [12.7 to 207.5]
  Cycle 2 - Days 19-20 (n=26, 28) | 23.15 [3.5 to 203.4] | 28.85 [3.5 to 159.3]
  Cycle 2 - Day 23 (n=27, 28) | 28.10 [3.5 to 159.3] | 32.15 [3.5 to 170.8]
  Cycle 2 - Day 24 (n=25, 28) | 36.80 [3.5 to 142.8] | 55.00 [3.5 to 200.0]
  Cycle 2 - Day 25 (n=27, 28) | 35.20 [3.5 to 148.5] | 62.30 [3.5 to 156.7]
  Cycle 2 - Day 27 (n=25, 28) | 39.60 [3.5 to 152.6] | 49.20 [3.5 to 127.6]
  Cycle 2 - Day 28 (n=26, 28) | 41.95 [3.5 to 149.8] | 55.05 [3.5 to 160.2]
  Cycle 3 - Day 2 (n=27, 28) | 54.70 [3.5 to 136.5] | 57.95 [3.5 to 162.3]
  Cycle 3 - Day 4 (n=27, 28) | 51.10 [3.5 to 122.1] | 52.25 [3.5 to 183.6]
  Cycle 3 - Day 6 (n=24, 26) | 36.15 [3.5 to 211.7] | 29.55 [3.5 to 141.4]
Statistical Analysis 1: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 2 time point. p-values < 0.05 were considered statistically significant; Test type: Superiority or Other; p = 0.0979, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 4 time point; Test type: Superiority or Other; p = 0.0629, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 6 time point; Test type: Superiority or Other; p = 0.8464, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Days 19-20 time point; Test type: Superiority or Other; p = 0.6316, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 23 time point; Test type: Superiority or Other; p = 0.3000, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 24 time point; Test type: Superiority or Other; p = 0.0955, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 25 time point; Test type: Superiority or Other; p = 0.1523, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 2 - Day 27 time point; Test type: Superiority or Other; p = 0.2809, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 28 time point; Test type: Superiority or Other; p = 0.8829, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 2 time point; Test type: Superiority or Other; p = 0.9262, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 -Day 4 time point; Test type: Superiority or Other; p = 0.7811, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: DR-1021 vs Mircette; Comparison of treatment groups at Cycle 3 - Day 6 time point; Test type: Superiority or Other; p = 0.3703, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Cycle 2 Days 1 - 20 to Cycle 2 Days 21 - 28 in Maximum Follicle Size
Description: The change in the size of the largest documented follicle during combination therapy (Days 1 to 21) and during monotherapy/placebo (Days 21-28) measured by trans-vaginal ultrasound.
Time Frame: Cycle 2, Days 1-20 and Cycle 2, Days 21-28
Population: Intent-to-treat population with available data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 18 | 18
mm | -2.02 (6.076) | -1.79 (3.081)

6. Secondary Outcome: Number of Days of Bleeding or Spotting During Unscheduled and Scheduled Study Periods
Description: The total number of days of unscheduled (Day 1 to Day 21 of each cycle) and scheduled (ie,withdrawal [Day 22 to Day 28 of each cycle]) bleeding or spotting was derived from participant diaries.
Time Frame: Cycle 2, Days 1-21, Cycle 2, Days 22-28 and Cycle 3, Days 1-21
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
days
  Cycle 2 - Unscheduled (Day 1-21) | 2.19 (3.732) | 1.41 (1.551)
  Cycle 2 - Scheduled (Day 22-28) | 3.19 (2.167) | 3.67 (1.754)
  Cycle 3 - Unscheduled (Day 1-21) | 1.96 (2.808) | 1.64 (2.614)

7. Secondary Outcome: Percentage of Participants With Bleeding or Spotting During Unscheduled and Scheduled Study Periods
Description: The percentage of participants with unscheduled (Day 1 to Day 21 of each cycle) and scheduled (ie,withdrawal [Day 22 to Day 28 of each cycle]) bleeding or spotting was derived from participant diaries.
Time Frame: Cycle 2, Days 1-21, Cycle 2, Days 22-28 and Cycle 3, Days 1-21
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
percentage of participants
  Cycle 2 - Unscheduled (Day 1-21) | 48.1 | 59.3
  Cycle 2 - Scheduled (Day 22-28) | 77.8 | 92.6
  Cycle 3 - Unscheduled (Day 1-21) | 55.6 | 53.6

8. Secondary Outcome: Number of Days of Bleeding During Unscheduled and Scheduled Study Periods
Description: The total number of days of unscheduled (Day 1 to Day 21 of each cycle) and scheduled (ie,withdrawal [Day 22 to Day 28 of each cycle]) bleeding (not including spotting) was derived from participant diaries.
Time Frame: Cycle 2, Days 1-21, Cycle 2, Days 22-28 and Cycle 3, Days 1-21
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
days
  Cycle 2 - Unscheduled (Day 1-21) | 0.70 (2.127) | 0.52 (0.935)
  Cycle 2 - Scheduled (Day 22-28) | 2.30 (1.793) | 2.63 (1.843)
  Cycle 3 - Unscheduled (Day 1-21) | 0.70 (1.436) | 0.71 (1.607)

9. Secondary Outcome: Percentage of Participants With Bleeding During Unscheduled and Scheduled Study Periods
Description: The percentage of participants with unscheduled (Day 1 to Day 21 of each cycle) and scheduled (ie,withdrawal [Day 22 to Day 28 of each cycle]) bleeding (not including spotting) was derived from participant diaries.
Time Frame: Cycle 2, Days 1-21, Cycle 2, Days 22-28 and Cycle 3, Days 1-21
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | DR-1021 | Mircette
Number analyzed (Participants) | 28 | 28
percentage of participants
  Cycle 2 - Unscheduled (Day 1-21) | 18.5 | 33.3
  Cycle 2 - Scheduled (Day 22-28) | 77.8 | 77.8
  Cycle 3 - Unscheduled (Day 1-21) | 29.6 | 25.0

ADVERSE EVENTS:
Time Frame: From the date of the first randomized dose through 14 days after the last randomized dose, up to 42 days.
Arm/Group | DR-1021 | Mircette
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/28
Other Adverse Events (participants affected / at risk) | 7/28 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-1021 (N=28) | Mircette (N=28)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-1021 (N=28) | Mircette (N=28)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.